CLINICAL TRIAL: NCT05172336
Title: Fetal Cardiac Remodeling in Singleton Pregnancies Conceived by Assisted Reproductive Technology (Biopsied and Non-Biopsied ICSI) Versus Those Normally Conceived
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wael Elbanna Clinic (Other)
Collaborators: National Research Centre, Egypt (Other)
Responsible Party: Sponsor
Other Study IDs: Elbanna_004
Record Dates: First submitted 2021-12-08; First posted 2021-12-29 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-08

CONDITIONS: Fetal Cardiac Disorder
Keywords: fetal echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Assisted reproductive technology (Biopsied ICSI): the study materials that will be used will include fetal ultrasound (fetal echocardiography) at 29 weeks ± 1week gestation.
- Assisted reproductive technology (Non-Biopsied ICSI): the study materials that will be used will include fetal ultrasound (fetal echocardiography) at 29 weeks ± 1week gestation.
- Spontaneous conception (SC): the study materials that will be used will include fetal ultrasound (fetal echocardiography) at 29 weeks ± 1week gestation.

SUMMARY:
The study aims to assess the presence of fetal cardiac remodeling and dysfunction in singleton pregnancies conceived by assisted reproductive technology (Biopsied and Non-Biopsied ICSI) as compared with those conceived spontaneously (SC).

DETAILED DESCRIPTION:
For gynecologists, reaching a conclusion about fetal cardiac remodeling and dysfunction in singleton pregnancies conceived by assisted reproductive technology (Biopsied and Non-Biopsied ICSI) or conceived spontaneously (SC) that would influence the clinical decision and best practice. Besides enriching the clinical evidence in fetal cardiac remodeling and dysfunction.

For society, the conclusion and recommendation shall maximize the benefits and managing the benefits of the technique used. Moreover, providing more information for fetal cardiac remodeling and dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged >18 years
2. Singleton pregnancy
3. Women who are willing and able to attend serial ultrasonographic examinations during the whole pregnancy
4. Women willing to sign an informed consent

Exclusion Criteria:

1. Multiple pregnancies; more than one fetus
2. Any maternal medical disease, including asthma, chronic hypertension, diabetes mellitus, heart disease, extracardiac anomalies, human immunodeficiency virus or hepatitis infection, immunological disorders, lupus, and thyroid disease
3. Diagnosis of fetal malformations; fetus with a structural or chromosomal anomaly
4. Fetus with Small-for-Gestational-Age (SGA) or intrauterine Growth Restriction (IUGR) (a fetal weight that is below the 10th percentile for gestational age) as determined through an ultrasound.
5. Smokers or drug/alcohol women
6. Inability to understand and provide written informed consent

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Singleton pregnant women conceived by:
  * Assisted reproductive technology (Biopsied ICSI)
  * Assisted reproductive technology (Non-Biopsied ICSI)
  * Spontaneous conception (SC)
Sampling Method: Non-Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2021-08-28 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
To assess the presence of fetal cardiac remodeling and dysfunction in singleton pregnancies conceived by assisted reproductive technology (Biopsied and Non-Biopsied ICSI) as compared with those conceived spontaneously (SC) | 2 weeks
  Recording the fetal echocardiography data including:
  1. Standard fetoplacental data
     * Estimated fetal weight (g)
     * Estimated fetal weight (centile)
     * Uterine artery mean PI
     * Umbilical artery PI
     * Middle cerebral artery PI
     * Cerebroplacental ratio
     * Ductus venosus PI
     * Aortic isthmus PI
  2. Cardiac morphometric data
     * Cardiothoracic ratio
     * Left atrial/heart ratio
     * Right atrial/heart ratio
     * Left ventricular sphericity index
     * Right ventricular sphericity index
     * Left ventricular free wall thickness (mm)
     * Septal wall thickness (mm)
     * Right ventricular free wall thickness (mm)
     * Myocardial Performance Index (MPI)
  3. Systolic function data
     * Left ejection fraction (%)
     * Right ejection fraction (%)
     * MAPSE (mm)
     * TAPSE (mm)
  4. Diastolic function data
     * Mitral E/A ratio
     * Tricuspid E/A ratio
     * Left isovolumic relaxation time (ms)
  5. Gestational age at ultrasound examination (weeks)

SECONDARY OUTCOMES:
To describe the baseline and perinatal characteristics in singleton fetuses conceived by assisted reproductive technology (Biopsied and Non-Biopsied ICSI) as compared with those conceived spontaneously (SC | 8 weeks
  1. Maternal characteristics
     * Age (years)
     * BMI (kg/m2)
     * Primiparous
  2. Pregnancy complications
     * Pre-eclampsia
     * Corticoid exposure
     * Gestational diabetes
  3. Delivery data
     * GA (weeks)
     * Cesarean section
     * Gender
     * Birth weight (g)
     * Birth weight centile
     * SGA (small-for gestational age)
  4. Neonatal outcome data
     * Admission to NICU
     * Major neonatal morbidity*

CONTACTS AND LOCATIONS:
Locations (1):
- National Research center, Cairo, Egypt